CLINICAL TRIAL: NCT04965883
Title: Comparison Between Early Excision and Grafting Versus Dressing and Delayed Grafting in Deep Burn Mangement.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shenoda Gamel Fayez, resident doctor at plastic surgery department sohag university hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Soh-Med-21-06-08
Record Dates: First submitted 2021-06-16; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Transplantation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Excision and Grafting (Experimental): * The early excision will be done surgically within 4-10 days post burn by whatson knife by tangential excision of burned tissue until capillary bleeding appears to make a good bed to be covered with grafts" split thickness grafts STG" at the same time.
  * The first dressing will be in the fifth day post operative.
  Interventions: Procedure: Excision and Grafting
- Dressing and Delayed Grafting (Experimental): • Dressing will be done for the second group every other day until spontanous eschar seperation or after surgiacl debridrment of adherent eschar then for delayed grafting more than 10 days post burn.
  Interventions: Procedure: dressing then delayed grafting

INTERVENTIONS:
Procedure: Excision and Grafting — reconstruction of deep burn by grafting
  Arms: Early Excision and Grafting
Procedure: dressing then delayed grafting — multiple dressing and delayed grafting
  Arms: Dressing and Delayed Grafting

SUMMARY:
* All the patients will be included in the study will be resuscitated on arrival in our department.
* Detailed history will be taken and burn evaluation will take place in respect to TBSA according to Lund and Browder chart and burn depth.
* Dreesing will be done with topical antimicrobial agent.
* Fluid resuscitation with lactated Ringer's solution according to modified Parkland's formula.
* Injectable proton pump inhibitors, and analgesics will be started as initial drug therapy.
* Close follow up of the patients will be done then evaluation of the patients will be done in the fourth day and dividing the patients into two groups: the first group "early exicion and grafting " and the second group " dressing and delayed grafting ".
* The first group will include patients with early surgery from 4 to 10 days since burn.
* Dressing will be done for the second group every other day until spontanous eschar seperation or after surgiacl debridrment of adherent eschar then for delayed grafting more than 10 days post burn.
* Then the data will be collected and analyzed for comparison between the two groups regarding : the timing of operation and its relation to the length of stay, functional outcome and cost of treatment

DETAILED DESCRIPTION:
* The first group will include :

  1. Patients with good general condition and hemodynamically stable that fit for early surgery.
  2. Patients that accept the option of early surgery and can give consent for it .
  3. Patients with available donor site for early grafting.
  4. Patients with burn at certain sites may be of priority for early excision and grafting to avoid long term complication of delayed wound healing such as : on joint surface, hands, feet, and face.
* The early excision will be done surgically within 4-10 days post burn by whatson knife by tangential excision of burned tissue until capillary bleeding appears to make a good bed to be covered with grafts" split thickness grafts STG" at the same time.
* The first dressing will be in the fifth day post operative.
* In the other hand the second group will include:

  1. Patients with bad general condition or hemodynamicaly unstable at the early excision period (4-10 days post burn).
  2. Patients that refuse early surgery and give no consent for early surgery.
  3. Patients with no available donner site for early excision and grafting during the fourth day evaluation .

ELIGIBILITY:
Inclusion Criteria:

1. Patients who had deep second and third degree burns.
2. patients with flame and scald burns.

Exclusion Criteria:

1. Patients who had only first or superficial second degree burns.
2. patients with high voltage contact electric burns and chemical burns.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-30 (Estimated); Primary Completion 2022-02-15 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Compare the number of blood units needed in both groups ( the first group : early exicion and grafting , the second group : dressing and delayed grafting ) | one year
  We will estimate how many blood units needed in both groups since admission upto discharge from hospital.
compare the cost of treatment in both groups | one year
  regarding how much money will be used since burn upto recovery measured by filling questionnaire by the patients.

SECONDARY OUTCOMES:
Compare the length of hospital stay between of early excision and grafting(EEG) versus dressing and delayed grafting(DDG) of deep burn. | one year
  how many days each group will spend in our hospital .

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Elmwalla, MD, Study Chair — Sohag university ,Egypt
Locations (1):
- Shenouda gamil fayiez, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forjuoh SN. Burns in low- and middle-income countries: a review of available literature on descriptive epidemiology, risk factors, treatment, and prevention. Burns. 2006 Aug;32(5):529-37. doi: 10.1016/j.burns.2006.04.002. Epub 2006 Jun 14. PMID 16777340
- [Background] Khadjibayev AM, Fayazov AD, Djabriyev DA, Kamilov UR. Surgical treatment of deep burns. Ann Burns Fire Disasters. 2008 Sep 30;21(3):150-2. PMID 21991128
- [Background] Janzekovic Z. A new concept in the early excision and immediate grafting of burns. J Trauma. 1970 Dec;10(12):1103-8. No abstract available. PMID 4921723